CLINICAL TRIAL: NCT04613531
Title: The Sensitivity and Specificity of Sniffer Dogs for Diagnosis of Parkinson's Disease: Diagnostic Accuracy Study
Brief Title: The Sensitivity and Specificity of Canine Detection of Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: Central South University (Other)
Collaborators: University of South China (Other); Mingji Hospital (Other)
Responsible Party: Principal Investigator, Chang-Qing Gao, Director, Center for studies in laboratory animals, Central South University
Other Study IDs: Xiang Ya 0005
Record Dates: First submitted 2020-10-28; First posted 2020-11-03 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples Without DNA — smell from participants' upper back
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants with PD: patients with clinically diagnosed Parkinson's disease
- Participants without PD: participants clinically diagnosed without Parkinsons' Disease

SUMMARY:
People sometimes report that their relatives who have been diagnosed with Parkinson's disease (PD) have a unique smell. A previous study has demonstrated that PD patients do have smell that is different from that of healthy people. Sniffer dogs have long been used to identify criminals, and recently been used to identify subject with cancer. The investigators hypothesized that sniffer dogs may be able to identify PD patients.

DETAILED DESCRIPTION:
Parkinson's Disease is a neurodegeneration disorder that affects the life of millions of people worldwide. There are multiple drugs available now that can modify the process of the disease. Making a timely and correct diagnosis of PD is still a great challenge in many cases even for specialists. Correct diagnosis is fundamental to the appropriate administration of medicines. To help clinicians to quickly and correctly make a diagnosis, the investigators aim to use sniffer dogs to identify PD patients from clearly non-PD subjects. After more than one-year training of the dogs, the investigators found that it is feasible to use dogs to identify PD patients from non-PD subjects. Now the investigators are trying to estimate the sensitivity and specificity of sniffer dogs in identifying PD patients from non-PD subjects.

In this multicenter study, the clinicians and their assistants will collect samples and send to the study center. One researcher alone will put seven plastic bags containing matched samples (one PD sample and six non-PD samples) on a table and take notes, then relabel them with random numbers and take notes again, and keep them in a confidential place till the study is completed. Another researcher will take over the relabeled samples and put them into different tanks and take notes. Thus, both the experimenter who helps to place the samples into tanks and the dog handler will not know the nature of the samples. Test results will be compared with the notes of the blind-setter after all the experiments have been performed. The sensitivity and specificity of identification will be calculated. The study aims to test the hypothesis that the diagnostic sensitivity of sniffer dogs in identifying PD patients from non-PD subjects is over 90%.

ELIGIBILITY:
Inclusion Criteria:

* Clinically established PD patients
* Clearly non-PD subjects will be recruited as controls

Exclusion Criteria:

* subjects with tremor or decrease of olfactory power or with rapid eye movement sleep behavior, obvious constipation, and depression.
* subjects who are taking antipsychotics.
* subjects with incomplete data.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: PD patients and other subjects in clinics
Sampling Method: Non-Probability Sample
Enrollment: 1198 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-01-22 (Actual); Study Completion 2021-01-22 (Actual)

PRIMARY OUTCOMES:
The specificity and sensitivity of the identification of PD patients from non-PD by at least 2 out of 3 sniffer dogs | Samples taken at the time of participant enrolment and assessed by the sniffer dogs within 20 weeks
  Sensitivity = number of samples of PD patients that were correctly identified by dogs/[number of samples of PD patients that were correctly identified+ number of samples of PD patients missed by the dogs]. One sample will be taken per patient.
  Specificity = number of samples of non-PD subjects that were correctly identified by dogs/[number of samples of non-PD subjects that were correctly identified by dogs + number of non-PD subjects that were identified as PD]. One sample will be taken per subject.

SECONDARY OUTCOMES:
Assess the accuracy of identification by sniffer dogs for PD patients with disease duration over five years and for those with disease duration within five years of diagnosis. | Samples taken at the time of participant enrolment and assessed by the sniffer dogs within 20 weeks
  Calculate sensitivity and specificity as mentioned above, but in two sub-populations: 1. PD patients with disease duration within 5 years and their control subjects; 2. PD patients with disease duration over 5 years and their control subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Chang-Qing Gao, MD,PhD, Study Director — Xiang-Ya Hospital, Central South University
Locations (1):
- XiangYa Hospital, Changsha, Hunan, China